CLINICAL TRIAL: NCT01969448
Title: A Prospective Randomized Trial to Assess Perfusion and Patient Satisfaction in Nipple-Areola Mastectomy With Immediate Reconstruction
Brief Title: Study to Assess Perfusion and Patient Satisfaction in Nipple-Areola Mastectomy With Immediate Reconstruction
Acronym: NASSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: LifeCell (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201302004
Record Dates: First submitted 2013-10-14; First posted 2013-10-25 (Estimated); Results first posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-03

CONDITIONS: Ductal Carcinoma in Situ - Category; Breast Cancer; Prophylactic Mastectomy
Keywords: Nipple-areola skin sparing mastectomy; Immediate reconstruction; Prophylactic Mastectomy; Breast-Q; Breast Cancer; Ductal Carcinoma in Situ - Category
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Inframammary Fold Incision Cohort (Active Comparator): * Inframammary fold incision which is in the crease under the breast.
  * Perfusion of the involved breast will be monitored at three separate time points using laser-assisted fluorescence angiography (Spy Elite, LifeCell)
    * Intraoperatively prior to mastectomy
    * At the conclusion of NASSM (following completion of mastectomy procedure and prior to implant insertion during reconstruction) - (ie. Mastectomy done, implant not in yet)
    * Following the conclusion of reconstruction with an immediate implant and skin closure with either temporary staples or final suture placement (ie. Mastectomy done and implant in)
  Interventions: Procedure: Inframammary Fold Incision; Device: Laser-assisted fluorescence angiography; Drug: Indocyanine Green
- Lateral Radial Incision Cohort (Active Comparator): * Lateral radial incision
  * Perfusion of the involved breast will be monitored at three separate time points using laser-assisted fluorescence angiography (Spy Elite, LifeCell)
    * Intraoperatively prior to mastectomy
    * At the conclusion of NASSM (following completion of mastectomy procedure and prior to implant insertion during reconstruction) - (ie. Mastectomy done, implant not in yet)
    * Following the conclusion of reconstruction with an immediate implant and skin closure with either temporary staples or final suture placement (ie. Mastectomy done and implant in)
  Interventions: Procedure: Lateral Radial Incision; Device: Laser-assisted fluorescence angiography; Drug: Indocyanine Green
- Non-Randomized Cohort (Other): * Patients in which the surgeon feels that for oncologic reasons must have a specific incision (either inframammary fold or lateral radial incision) and cannot be randomized due to concerns of compromising clinical care but otherwise meet the inclusion and exclusion criteria will be offered participation as part of a non-randomized cohort.
  * Perfusion of the involved breast will be monitored at three separate time points using laser-assisted fluorescence angiography (Spy Elite, LifeCell)
    * Intraoperatively prior to mastectomy
    * At the conclusion of NASSM (following completion of mastectomy procedure and prior to implant insertion during reconstruction) - (ie. Mastectomy done, implant not in yet)
    * Following the conclusion of reconstruction with an immediate implant and skin closure with either temporary staples or final suture placement (ie. Mastectomy done and implant in)
  Interventions: Procedure: Inframammary Fold Incision or Lateral Radial Incision; Device: Laser-assisted fluorescence angiography; Drug: Indocyanine Green

INTERVENTIONS:
Procedure: Inframammary Fold Incision or Lateral Radial Incision
  Arms: Non-Randomized Cohort
Procedure: Lateral Radial Incision
  Arms: Lateral Radial Incision Cohort
Procedure: Inframammary Fold Incision
  Arms: Inframammary Fold Incision Cohort
Device: Laser-assisted fluorescence angiography
  Other Names: Spy Elite, LifeCell.
Drug: Indocyanine Green

SUMMARY:
The investigators hypothesize that nipple-areola skin sparing mastectomy (NASSM) performed through an inframammary incision has a superior blood supply relative to a lateral oblique incision. Moreover, by minimizing complications and optimizing aesthetic outcomes, the investigators believe it will be associated with significantly higher patient reported outcome scores. The addition of information gained by use of intraoperative laser-assisted fluorescent angiography (measured with the Spy Elite imaging device) will reduce complication rates by directing intraoperative resection of ischemic tissue and limiting the volume of immediate implant placement in instances where real time imaging would suggest compromised perfusion. These quantifiable, objective measures will justify the use of NASSM and immediate implant placement coupled with intraoperative laser-assisted fluorescent angiography in prosthetic based breast reconstruction despite longer operative times.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be scheduled to undergo either a single or bilateral elective nipple-areola skin sparing mastectomy (NASSM) procedure with planned immediate reconstruction.
* Patient must be 18 years of age or older.
* Karnofsky Performance Scale of at least 80%.
* Patient must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Cognitive impairment.
* BMI < 18 or > 35
* Breast >800 grams or <100 grams in predicted weight. "Breast" includes the breast tissue and in cases where the patient already has cosmetic breast implants, the additional breast implant mass. The sum total must be >100 g and <800 g.
* History of radiation to the chest wall or breast being studied
* Patients who have a history of allergy to iodides or iodinated contrast agents
* Surgeon's opinion at the time of surgery that the subject's well-being would be compromised (e.g. significant comorbidities, intraoperative findings of a higher stage cancer or other independent acute health problems). If the contralateral breast is undergoing a nipple-sparing mastectomy with reconstruction as well, then the contralateral breast can be studied so long as there is no compromise to any element of their care.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-03-28 (Actual); Primary Completion 2016-04-27 (Actual); Study Completion 2017-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marissa J Tenenbaum, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim HJ, Park EH, Lim WS, Seo JY, Koh BS, Lee TJ, Eom JS, Lee SW, Son BH, Lee JW, Ahn SH. Nipple areola skin-sparing mastectomy with immediate transverse rectus abdominis musculocutaneous flap reconstruction is an oncologically safe procedure: a single center study. Ann Surg. 2010 Mar;251(3):493-8. doi: 10.1097/SLA.0b013e3181c5dc4e. PMID 20134317
- [Background] Cense HA, Rutgers EJ, Lopes Cardozo M, Van Lanschot JJ. Nipple-sparing mastectomy in breast cancer: a viable option? Eur J Surg Oncol. 2001 Sep;27(6):521-6. doi: 10.1053/ejso.2001.1130. PMID 11520082
- [Background] Paepke S, Schmid R, Fleckner S, Paepke D, Niemeyer M, Schmalfeldt B, Jacobs VR, Kiechle M. Subcutaneous mastectomy with conservation of the nipple-areola skin: broadening the indications. Ann Surg. 2009 Aug;250(2):288-92. doi: 10.1097/SLA.0b013e3181b0c7d8. PMID 19638905
- [Background] de Alcantara Filho P, Capko D, Barry JM, Morrow M, Pusic A, Sacchini VS. Nipple-sparing mastectomy for breast cancer and risk-reducing surgery: the Memorial Sloan-Kettering Cancer Center experience. Ann Surg Oncol. 2011 Oct;18(11):3117-22. doi: 10.1245/s10434-011-1974-y. Epub 2011 Aug 17. PMID 21847697
- [Background] Salzberg CA, Ashikari AY, Koch RM, Chabner-Thompson E. An 8-year experience of direct-to-implant immediate breast reconstruction using human acellular dermal matrix (AlloDerm). Plast Reconstr Surg. 2011 Feb;127(2):514-524. doi: 10.1097/PRS.0b013e318200a961. PMID 21285756
- [Background] Sacchini V, Pinotti JA, Barros AC, Luini A, Pluchinotta A, Pinotti M, Boratto MG, Ricci MD, Ruiz CA, Nisida AC, Veronesi P, Petit J, Arnone P, Bassi F, Disa JJ, Garcia-Etienne CA, Borgen PI. Nipple-sparing mastectomy for breast cancer and risk reduction: oncologic or technical problem? J Am Coll Surg. 2006 Nov;203(5):704-14. doi: 10.1016/j.jamcollsurg.2006.07.015. Epub 2006 Sep 11. PMID 17084333
- [Background] Palmieri B, Baitchev G, Grappolini S, Costa A, Benuzzi G. Delayed nipple-sparing modified subcutaneous mastectomy: rationale and technique. Breast J. 2005 May-Jun;11(3):173-8. doi: 10.1111/j.1075-122X.2005.21520.x. PMID 15871701
- [Background] Gerber B, Krause A, Dieterich M, Kundt G, Reimer T. The oncological safety of skin sparing mastectomy with conservation of the nipple-areola complex and autologous reconstruction: an extended follow-up study. Ann Surg. 2009 Mar;249(3):461-8. doi: 10.1097/SLA.0b013e31819a044f. PMID 19247035
- [Background] Tepper OM, Karp NS, Small K, Unger J, Rudolph L, Pritchard A, Choi M. Three-dimensional imaging provides valuable clinical data to aid in unilateral tissue expander-implant breast reconstruction. Breast J. 2008 Nov-Dec;14(6):543-50. doi: 10.1111/j.1524-4741.2008.00645.x. PMID 19054001
- [Background] Lista F, Ahmad J. Vertical scar reduction mammaplasty: a 15-year experience including a review of 250 consecutive cases. Plast Reconstr Surg. 2006 Jun;117(7):2152-65; discussion 2166-9. doi: 10.1097/01.prs.0000218173.16272.6c. PMID 16772910
- [Background] Garwood ER, Moore D, Ewing C, Hwang ES, Alvarado M, Foster RD, Esserman LJ. Total skin-sparing mastectomy: complications and local recurrence rates in 2 cohorts of patients. Ann Surg. 2009 Jan;249(1):26-32. doi: 10.1097/SLA.0b013e31818e41a7. PMID 19106672
- [Background] Ashikari RH, Ashikari AY, Kelemen PR, Salzberg CA. Subcutaneous mastectomy and immediate reconstruction for prevention of breast cancer for high-risk patients. Breast Cancer. 2008;15(3):185-91. doi: 10.1007/s12282-008-0059-7. PMID 18575951
- [Background] Gerber B, Krause A, Reimer T, Muller H, Kuchenmeister I, Makovitzky J, Kundt G, Friese K. Skin-sparing mastectomy with conservation of the nipple-areola complex and autologous reconstruction is an oncologically safe procedure. Ann Surg. 2003 Jul;238(1):120-7. doi: 10.1097/01.SLA.0000077922.38307.cd. PMID 12832974
- [Background] Komorowska-Timek E, Gurtner GC. Intraoperative perfusion mapping with laser-assisted indocyanine green imaging can predict and prevent complications in immediate breast reconstruction. Plast Reconstr Surg. 2010 Apr;125(4):1065-1073. doi: 10.1097/PRS.0b013e3181d17f80. PMID 20335859
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Losken A, Zenn MR, Hammel JA, Walsh MW, Carlson GW. Assessment of zonal perfusion using intraoperative angiography during abdominal flap breast reconstruction. Plast Reconstr Surg. 2012 Apr;129(4):618e-624e. doi: 10.1097/PRS.0b013e3182450b16. PMID 22456376
- [Background] Ashitate Y, Lee BT, Ngo LH, Laurence RG, Hutteman M, Oketokoun R, Lunsford E, Soo Choi H, Frangioni JV. Quantitative assessment of nipple perfusion with near-infrared fluorescence imaging. Ann Plast Surg. 2013 Feb;70(2):149-53. doi: 10.1097/SAP.0b013e31822f9af7. PMID 21862913
- [Derived] Odom EB, Parikh RP, Um G, Kantola SW, Cyr AE, Margenthaler JA, Tenenbaum MM, Myckatyn TM. Nipple-Sparing Mastectomy Incisions for Cancer Extirpation Prospective Cohort Trial: Perfusion, Complications, and Patient Outcomes. Plast Reconstr Surg. 2018 Jul;142(1):13-26. doi: 10.1097/PRS.0000000000004498. PMID 29878989
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment to the study opened to enrollment 03/28/2013 and closed to enrollment on 03/09/2016.
Period: Overall Study
Arm/Group | Inframammary Fold Incision Cohort | Lateral Radial Incision Cohort | Non-Randomized Cohort
Started | 55 | 24 | 0
Completed | 55 | 24 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inframammary Fold Incision Cohort | Lateral Radial Incision Cohort | Non-Randomized Cohort | Total
Number analyzed (Participants) | 55 | 24 | 0 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (10.8) | 46.6 (10.5) |  | 44.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 24 | 0 | 79
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 55 | 24 |  | 79

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Original Preoperative Blood Supply (Perfusion) Post Nipple Sparing Mastectomy
Description: * Laser-assisted fluorescent angiography via the Spy Elite imaging device will be utilized to capture this data during mastectomy and immediate breast reconstruction. Standard postoperative patient follow up will assess for perfusion.
  * The Spy device quantifies perfusion by measuring relative fluorescence of indocyanine green bound to plasma proteins. This produces an intensity value of 0-255 based on an 8-bit greyscale. The investigators measured this value preoperatively when measured and compared to the post-intervention measurement. The device can calculate the cumulative intensity of a defined region of interest which the investigators categorized as the lateral, lower, medial, or nipple-areola region of the breast. The investigators also evaluated the cumulative value of these areas in total. Rate of perfusion was simply this value over time (90 seconds).
Time Frame: At the time of surgery (day 1)
Measure: Number; unit: percentage of original preop perfusion
Arm/Group | Inframammary Fold Incision Cohort | Lateral Radial Incision Cohort | Non-Randomized Cohort
Number analyzed (Participants) | 55 | 24 | 0
percentage of original preop perfusion
  Overall breast | 63.9 | 60.8 |
  Nipple | 29.9 | 40.0 |
  Inferior | 54.6 | 72.0 |
  Lateral | 73.5 | 76.5 |
  Medial | 62.5 | 65.2 |

2. Primary Outcome: Percentage of Original Preoperative Blood Supply (Perfusion) Post Reconstruction
Description: as for outcome 1
Time Frame: At the time of surgery (day 1)
Measure: Number; unit: percentage of original preop perfusion
Arm/Group | Inframammary Fold Incision Cohort | Lateral Radial Incision Cohort | Non-Randomized Cohort
Number analyzed (Participants) | 55 | 24 | 0
percentage of original preop perfusion
  Overall breast | 30.6 | 35.1 |
  Nipple | 23.2 | 31.3 |
  Inferior | 21.9 | 36.9 |
  Lateral | 23.01 | 40.7 |
  Medial | 28.0 | 32.1 |

3. Secondary Outcome: Breast Q Score
Description: -The BREAST-Q is a previously validated instrument which measures patient reported outcomes. It has several iterations including the one utilized here which is specific for implant-based breast reconstruction. Each of its 6 domains generates a Q-score from 0 (lowest) to 100 (highest). A higher number indicates a higher satisfaction or better quality of life than a lower number. Based on answers to the questions, each individual will generate a whole number score for each domain. The patient can be sampled preoperatively and postoperatively as well as over time to calculate the impact of intervention and time on this value. Q-scores are calculated for each domain, and the investigators report a mean value based on data from an entire cohort for the particular domain. Domains include evaluation of overall satisfaction with breasts, physical well being, sexual well being, as well as satisfaction with office staff, information provided, and the provider.
Time Frame: Up to 3 months post permanent implant placement
Population: 6 participants were not evaluable for this outcome measure in the inframammary fold incision cohort and 2 particpants were not evaluable for this outcome measure in the lateral radial incision cohort due to not completing the Breast Q score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inframammary Fold Incision Cohort | Lateral Radial Incision Cohort | Non-Randomized Cohort
Number analyzed (Participants) | 49 | 22 | 0
units on a scale
  Satisfaction with Breasts (pre-op) | 62.1 (17.3) | 53.8 (13.1) |
  Satisfaction with Breasts (post-op) | 69.3 (21.8) | 68.7 (12.0) |
  Psychosocial (pre-op) | 74.1 (16.5) | 68.0 (12.9) |
  Psychosocial (post-op) | 79.8 (19.8) | 85.2 (17.0) |
  Physical chest (pre-op) | 88.3 (14.0) | 85.7 (12.2) |
  Physical chest (post-op) | 77.9 (12.4) | 83.4 (12.4) |
  Sexuality (pre-op) | 59.4 (10.3) | 56.7 (10.8) |
  Sexuality (post-op) | 68.7 (25.3) | 68.6 (17.2) |

4. Secondary Outcome: Number of Participants With Tissue Expander
Time Frame: Up to 3 months post permanent implant placement
Measure: Count of Participants; unit: Participants
Arm/Group | Inframammary Fold Incision Cohort | Lateral Radial Incision Cohort | Non-Randomized Cohort
Number analyzed (Participants) | 55 | 24 | 0
Participants | 19 | 12 |

5. Secondary Outcome: Mean Operative Times for Mastectomy
Time Frame: At the time of surgery (day 1)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Inframammary Fold Incision Cohort | Lateral Radial Incision Cohort | Non-Randomized Cohort
Number analyzed (Participants) | 55 | 24 | 0
minutes | 155.3 (41.2) | 177.0 (29.0) |

6. Secondary Outcome: Breast Weight
Time Frame: At time of surgery (day 1)
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Inframammary Fold Incision Cohort | Lateral Radial Incision Cohort | Non-Randomized Cohort
Number analyzed (Participants) | 55 | 24 | 0
grams | 350 (156) | 418 (151) |

ADVERSE EVENTS:
Description: Common complications occur with breast oncologic and reconstructive surgery. None of these are expected to be related to the performance of this study and will not be summarized, graded or reported as traditional adverse event reporting in an interventional oncology trial.
Arm/Group | Inframammary Fold Incision Cohort | Lateral Radial Incision Cohort | Non-Randomized Cohort
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/24 | 0/0
Other Adverse Events (participants affected / at risk) | 0/55 | 0/24 | 0/0

LIMITATIONS AND CAVEATS:
Study had randomized-controlled trial design with assignment to IMF or LR incision but during enrollment patients frequently withdrew from randomization due to patient/surgical oncology preference and/or preexisting scars precluding randomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes